CLINICAL TRIAL: NCT01577875
Title: A Prospective Clinical Study to Evaluate Narrow Band Imaging and Magnifying Colonoscopy for the Histologic Prediction of Colorectal Polyps
Brief Title: Comparison of Narrow Band Imaging With or Without Magnifying Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NBI_Zoom_CVS_01
Record Dates: First submitted 2012-04-10; First posted 2012-04-16 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2012-04

CONDITIONS: Intestinal Polyps
MeSH Terms: conditions — Intestinal Polyps | interventions — Narrow Band Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): histologic prediction only with the narrow band imaging (without magnification)
- test group (Other): histologic prediction with narrow band imaging plus magnification
  Interventions: Device: NBI with magnification

INTERVENTIONS:
Device: NBI with magnification — After randomization of the subjects into two groups(1) NBI with magnification, 2) without magnification), one experienced endoscopist records its site, size, shape, and predicted histologic diagnosis on the every polyp observed and endoscopically resected. Two groups will be compared with each other.
  Other Names: Narrow band image with magnification
  Arms: test group

SUMMARY:
The aim of this study is to evaluate the usefulness of magnifying colonoscopy with narrow band imaging.

DETAILED DESCRIPTION:
The accuracy of histologic prediction for the colorectal polyps with the use of narrow band imaging is evaluated between the test group with magnifying colonoscopy and the control group without magnifying colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with colorectal polyps which are in need of EMR

Exclusion Criteria:

* pregnancy, IBD, colorectal cancer, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Accuracy of colorectal polyp histologic prediction with NBI colonoscopy plus magnification | After 1 week
  After radomization of the subjects into two groups(1) NBI with magnification, 2) without magnification), one experienced endoscopist records its site, size, shape, and predicted histologic diagnosis on the every polyp observed and endoscopically resected. After 1 week, confirmed pathologic diagnosis and predicted histologic diagnosis based on endoscopic observation are compared and its accuracy is evaluated.

SECONDARY OUTCOMES:
Sensitivity of the endoscopic histologic prediction with NBI plus magnification | 1 Week
  Endoscopically predicted histologic diagnosis compared with confirmed pathologic diagnosis are evaluated in terms of sensitivity.
Specificity of the endoscopic histologic prediction with NBI plus magnification | 1 Week
  Endoscopically predicted histologic diagnosis compared with confirmed pathologic diagnosis are evaluated in terms of specificity.
Positive predictive value of the endoscopic histologic prediction with NBI plus magnification | 1 Week
  Endoscopically predicted histologic diagnosis compared with confirmed pathologic diagnosis are evaluated in terms of positive predictive value.
Negative predictive value of the endoscopic histologic prediction with NBI plus magnification | 1 Week
  Endoscopically predicted histologic diagnosis compared with confirmed pathologic diagnosis are evaluated in terms of negative predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Sup Hong, MD, Principal Investigator — SNUH Internal Medicine
Locations (1):
- SNUH, Jongno-gu, Seoul, South Korea